CLINICAL TRIAL: NCT04081740
Title: Biological Determinants of Sputum Rheology in Chronic Airway Diseases
Acronym: CADRhé
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: APARD Fonds de dotation (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0430
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Asthma; COPD; Bronchiectasis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthma: The patients included in this group will have asthma, as specified in the inclusion criteria.
- COPD: The patients included in this group will have COPD, as specified in the inclusion criteria.
- Bronchiectasis: The patients included in this group will have bronchiectasis, as specified in the inclusion criteria.

SUMMARY:
The primary objective of this study is to investigate the biological determinants of sputum rheology variations.

DETAILED DESCRIPTION:
Secondarily, this study aims to compare rheology parameters between different chronic airway disease sub-populations.

ELIGIBILITY:
Inclusion Criteria:

* Affiliate with or beneficiary of the French national single-payer health insurance system
* Patient capable of spontaneous mucus expectoration
* Consulting or hospitalized at the study centre

Inclusion Criteria for the Asthma Group

* Never- or former-smoker (<10 pack-years)
* Medical history compatible with asthma
* Reversible post-brochodilator (or post-corticosteroid test) ventilatory obstruction (ratio of forced expiratory volume in 1 second : forced vital capacity < 70%) or significant variation in respiratory function -- OR -- Bronchial hyperresponsiveness demonstrated during a broncho-provocation test

Inclusion Criteria for the COPD Group

* Current- or former-smokers (>10 pack years)
* Chronic obstructive pulmonary disease according to GOLD criteria

Inclusion Criteria for the Bronchiectasis Group

* Presence of bronchiectasis on computed tomography scan
* Cystic fibrosis has been ruled out

Exclusion Criteria:

* Patient expresses opposition to the protocol
* Breast feeding or pregnant
* Metastatic neoplastic disease
* Other active pulmonary disease (tuberculosis, interstitial lung disease)
* Recent psychiatric disorder (in the past year and documented via a specialist consult)
* Consumption of illicit drugs or alcoholism
* Patients in an exclusion period determined by another study
* Patients under any type of legal guardianship
* Prisoners
* Impossible to correctly inform the patient
* Does not fluently read French
* Emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to patients with a chronic airway disease (asthma, chronic obstructive pulmonary disease (COPD) or bronchiectasis) present at the study centre and capable of spontaneous mucus expectoration.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Measurement of crossover stress (mucus rheology) | Day 0
  The crossover stress point for each mucus sample will be measured in Pa.

SECONDARY OUTCOMES:
Measurement of the storage modulus (mucus rheology) | Day 0
  The storage modulus point for each mucus sample will be measured in Pa.
Measurement of the loss modulus (mucus rheology) | Day 0
  The loss modulus point for each mucus sample will be measured in Pa.
Measurement of the strain crossover (mucus rheology) | Day 0
  The strain crossover point for each mucus sample will be measured in Pa.
Measurement of the loss factor (mucus rheology) | Day 0
  The loss factor point for each mucus sample will be measured as a tangent to an angle in radians.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Volpato, MS, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Arnaud de Villeneuve Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to, in as much as possible, make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity. Due to conditions imposed by French law, data will be made available to the public upon request to the study sponsor and fulfilment of French legal requirements.
Time Frame: Requests for individual datasets can be made anytime following full publication of results.
Access Criteria: Due to French law there are restrictions on publicly sharing the data of this study. Data requests may be submitted to the study sponsor and must be approved by the French data protection authority (la Commission Nationale de l'Informatique et des Libertés (CNIL)). French law requires that everyone who wishes to access clinical study data on humans must ask the CNIL for permission. For further information, please see: https://www.cnil.fr/.

REFERENCES:
- [Derived] Volpato M, Vialaret J, Hirtz C, Petit A, Suehs C, Patarin J, Matzner-Lober E, Vachier I, Molinari N, Bourdin A, Charriot J. Rheology predicts sputum eosinophilia in patients with muco-obstructive lung diseases. Biochem Biophys Res Commun. 2022 Sep 24;622:64-71. doi: 10.1016/j.bbrc.2022.07.025. Epub 2022 Jul 11. PMID 35843096